CLINICAL TRIAL: NCT00358306
Title: The Role of Endothelium Dysfunction in Progression of CKD (Chronic Kidney Disease) After AKI (Acute Kidney Injury)
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, David Askenazi, Principal Investigator, University of Alabama at Birmingham
Other Study IDs: F070309010
Record Dates: First submitted 2006-07-28; First posted 2006-07-31 (Estimated); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Acute Renal Failure; Chronic Kidney Failure; Endothelial Dysfunction; Hemolytic-uremic Syndrome (HUS)
Keywords: Endothelium; Chronic Kidney Disease; Acute Kidney Injury; Hemolytic-uremic syndrome (HUS)
MeSH Terms: conditions — Acute Kidney Injury; Kidney Failure, Chronic; Hemolytic-Uremic Syndrome; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- a: those with previous history of Acute kidney injury

SUMMARY:
To understand how AKI (Acute Kidney Injury) leads to chronic kidney disease so therapies can be found to alter the progression of events thereby significantly impacting the long-term outcomes of children who develop AKI.

DETAILED DESCRIPTION:
This research study is designed to study what happens to the kidneys after they have an injury. There is some evidence that even if there appears to be great improvement of kidney function, an injury can put patients at risk for long-term problems with their kidney function and increase their risk to have high blood pressure. We want to collect information from participants to help explain why this injury can cause future problems, including Chronic Kidney Disease (CKD) which may help us prevent these health problems.

ELIGIBILITY:
Inclusion Criteria:

* Children between age 2-20
* Decrease in renal function by 25% or greater
* Renal function has returned to normal

Exclusion Criteria:

* History of chronic disease
* Cancer
* Congenital heart disease
* Organ Transplantation
* Liver disease
* Pulmonary disease
* Diabetes other primary metabolic condition
* Severe neurologic impairments
* Hypertension
* Auto-immune
* Infectious disease or renal disease
* Smokers
* Renal disease w/primary cause i.e. - HUS or Glomerulonephritis
* severe allergies including allergy to seafood and/or iodine

Ages: 2 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children 2-20 years old with history of acute kidney injury
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2008-04; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Askenazi, MD, Principal Investigator — UAB Pediatric Nephrology
Locations (1):
- University Of Alabama, Birmingham, Alabama, United States